CLINICAL TRIAL: NCT06351592
Title: First in Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Ascending Doses of Intrathecally Administered ALN-SOD in Participants With Amyotrophic Lateral Sclerosis and SOD1 Mutations
Brief Title: First in Human (FIH) Study of ALN-SOD in Adult Participants With Amyotrophic Lateral Sclerosis Associated With Mutation in the SOD1 Gene (SOD1-ALS)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-SOD-ALS-2351; 2023-510344-20-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Mutation in the Superoxide Dismutase-1 (SOD1) Gene
Keywords: Symptomatic; Known pathogenic mutation; Predicted pathogenic mutation
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No masking during Open-Label Treatment Period after 4-week Double-Blind Treatment Period. This part of the study consists of a crossover design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Cohort 1 - Low Dose (Experimental): Placebo during double-blind treatment period
  Interventions: Drug: ALN-SOD; Other: Diluent; Drug: Placebo (PB)
- Cohort 2 - Mid Dose (Experimental): Placebo during double-blind treatment period
  Interventions: Drug: ALN-SOD; Other: Diluent; Drug: Placebo (PB)
- Cohort 3 - High Dose (Experimental): Placebo during double-blind treatment period
  Interventions: Drug: ALN-SOD; Other: Diluent; Drug: Placebo (PB)
- Cohort 4 (Optional) ≤ High Dose (Experimental): Placebo during double-blind treatment period
  Interventions: Drug: ALN-SOD; Other: Diluent; Drug: Placebo (PB)

INTERVENTIONS:
Drug: ALN-SOD — Administered by intrathecal (IT) injection
Other: Diluent — Administered by IT injection
Drug: Placebo (PB) — Administered by IT injection

SUMMARY:
This study is researching an experimental drug called ALN-SOD (called "study drug"). This study is focused on people with amyotrophic lateral sclerosis (ALS) caused by a change in a gene called the superoxide dismutase-1 (SOD1) gene. This type of ALS is known as "SOD1-ALS". This is the first time that ALN-SOD will be given to people. The aim of the study is to see how safe and tolerable the study drug is.

The study is looking at several other research questions, including:

* The effect the study drug has on specific biomarkers, which are substances in the blood or in the fluid that surrounds the brain and spinal cord, known as cerebrospinal fluid (CSF)
* How much study drug is in the blood and in the CSF, at different times
* Whether the body makes antibodies against the study drug (which could make the drug less effective or could lead to side effects)
* What effects the study drug has on ALS symptoms

ELIGIBILITY:
Key Inclusion Criteria:

1. Weakness attributable to ALS and a SOD1 mutation that has been previously described as associated with ALS or is considered likely to cause ALS, as defined in the protocol
2. Slow vital capacity (SVC) ≥50% predicted value based on age, gender and height, measured in upright position
3. Body Mass Index (BMI) ≤35 kg/m2 at time of screening
4. If participants are taking riluzole or edaravone, they must be on a stable dose for at least 4 weeks prior to initial dosing visit and are expected to remain at that dose until the end of the study
5. Platelet count >50,000/microliter
6. Has normal blood pressure readings, as defined in the protocol

Key Exclusion Criteria:

1. Concurrent participation in another interventional clinical trial
2. Has had a tracheostomy
3. Has dementia, as assessed by the investigator
4. Has uncontrolled psychiatric disease, including psychosis, active or recent suicidal ideation, untreated major depression, in the past 30 days
5. Has a medical history of brain or spinal disease/injury that would interfere with the lumbar puncture (LP) process, CSF circulation or safety assessment, as defined in the protocol
6. Presence of an implanted shunt for the drainage of CSF or an implanted central nervous system (CNS) catheter
7. Presents any concern to the study investigator that might confound the results of the study or poses an additional risk to the participant by their participation in the study
8. Was hospitalized (ie, >24 hours) for any reason other than ALS within 30 days of screening
9. Has received treatment with tofersen within 6 months prior to screening

NOTE: Other protocol defined inclusion / exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2029-04-26 (Estimated); Study Completion 2029-04-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse event (TEAEs) in participants treated with ALN-SOD | At week 4 and week 124
Severity of TEAEs in participants treated with ALN-SOD | At week 4 and week 124

SECONDARY OUTCOMES:
Concentration of neurofilament light chain (NfL) in plasma over time | Up to approximately week 124
Change in concentration of NfL in plasma over time | Up to approximately week 124
Concentration of SOD1 protein in cerebrospinal fluid (CSF) over time | Up to approximately week 124
Change in concentration of SOD1 protein in CSF over time | Up to approximately week 124
Concentration of NfL in CSF over time | Up to approximately week 124
Change in concentration of NfL in CSF over time | Up to approximately week 124
Change in Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) over time | Up to approximately week 124
Concentration of ALN-SOD in plasma over time | Up to approximately week 124
Concentration of ALN-SOD in CSF over time | Up to approximately week 124
Incidence of anti-drug antibodies (ADAs) to ALN-SOD in serum over time | Up to approximately week 124
Titer of ADAs to ALN-SOD in serum over time | Up to approximately week 124

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (14):
- Australia (3):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Sunshine Coast University Hospital, Birtinya, Queensland
- Canada (4):
  - University of Alberta Hospital, Edmonton, Division of Neurology, Edmonton, Alberta
  - University Hospital - London Health Sciences Centre, London, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Japan (4):
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Tokushima University Hospital, Tokushima, Tokushima
  - Toho University Omori Medical Center, Ōta-ku, Tokyo
  - Kyoto University Hospital, Kyoto
- South Korea (2):
  - Hanyang University Seoul Hospital, Seoul
  - Seoul National University Hospital, Seoul
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued development of the product for all indications on or after April 2020 and has no plans for future development
  * made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/